CLINICAL TRIAL: NCT03544073
Title: Does a GnRH Agonist Given at Embryo Transfer Improve Clinical Pregnancy and Live Birth Rates of Women Undergoing In-Vitro Fertilization?
Brief Title: GnRH Agonist at Embryo Transfer: IVF Outcomes
Acronym: GRAET
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The investigators were not able to get grant funding for this study.
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-03-14
Record Dates: First submitted 2018-05-21; First posted 2018-06-01 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Infertility; Infertility, Female; Infertility, Male
Keywords: in-vitro fertilization
MeSH Terms: conditions — Infertility; Infertility, Female; Infertility, Male | interventions — Saline Solution; Injections; Leuprolide

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Patient and provider will both be blinded to the medication that the patient receives.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Saline Solution for Injection (Placebo Comparator): This arm will receive a one-time subcutaneous injection of 0.4mL normal saline solution at the time of embryo transfer. This arm will continue to receive all the same treatments that everyone routinely receives for the IVF cycle, e.g. estrogen and progesterone supplements.
  Interventions: Drug: Saline Solution for Injection
- Leuprolide Acetate (Experimental): This arm will receive a one-time subcutaneous injection of 0.4U (0.2mg=0.4mL) Leuprolide acetate at the time of embryo transfer. This arm will continue to receive all the same routine treatments for the IVF cycle, e.g. estrogen and progesterone supplements.
  Interventions: Drug: Leuprolide Acetate

INTERVENTIONS:
Drug: Saline Solution for Injection — Placebo arm will receive a saline injection
  Other Names: NS; NSS
  Arms: Saline Solution for Injection
Drug: Leuprolide Acetate — Treatment arm will receive a Leuprolide injection
  Other Names: Lupron
  Arms: Leuprolide Acetate

SUMMARY:
In ART (assisted reproductive technology) cycles, embryos are transferred to a woman's uterus after in-vitro fertilization (IVF) in a laboratory. Usually, hormones (progesterone) are given to the patient after transferring the embryo, as a supplement, in order to mimic the natural hormones that would normally be secreted in an unassisted pregnancy. This study will identify whether additional gonadotropin-releasing hormone (GnRH-agonist) administration, a natural hormone secreted from the hypothalamus, will improve the clinical pregnancy and live birth rates when using IVF.

DETAILED DESCRIPTION:
This is a randomized, double-blinded, placebo-controlled study. On the day of embryo transfer (5-6 days after a fresh egg retrieval and on the 6th day of progesterone administration in a frozen embryo transfer cycle), patients will receive either a single injection of 20 Units (1mg) of Lupron or an identical placebo injection. Patients undergoing day 3 embryo transfers will not be eligible and will not be randomized.

Randomization will be in 22 blocks of 20 patients. Based on the power analysis with a power of 0.8 and alpha-error of 0.05, the investigators will need to enroll 352 patients, so the investigators will recruit 440 to account for attrition.

Randomization scheme will be computed via a computerized program accessible at randomization.com or via SPSS. There will be one randomization: both fresh and frozen embryo cycles will be randomized in the same group. Sequential cards with randomization allocation will be placed in doubly sealed, opaque envelopes, with a single sheet confirming eligibility status. Confirmation of the presence of the signed Informed Consent will be in the first envelope. The second envelope will be opened after there is confirmation that the patient is eligible and consented. This envelope will have a card stating the group the patient has been assigned to, with blank spaces designated to record patient information. This card will be completed by the study staff and saved for reference purposes. The card will state the group that the patient was randomized to, the date of embryo transfer, the patient's medical record number, name, and cycle type. There will also be a log book to record the information and medication lot numbers.

Injections will be prepared at the time of randomization by the research coordinator and will be administered by the clinical RN, who will not know its contents. The clinical staff assessing and planning care of the patient (attending physicians and nurses) will not know the contents of the syringe (either Lupron 20 IU or the same amount of normal saline).

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing in-vitro fertilization who are receiving an embryo transfer of a day 5 blastocyst

Exclusion Criteria:

* Those who have a contraindication to receiving the medication

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-15 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | 2 years
  Percentage of live births for all patients included.

SECONDARY OUTCOMES:
Miscarriage rate | 2 years
  Percentage of pregnancies that ended in miscarriage
Clinical pregnancy rate | 2 years
  Percentage of patients who had a clinical pregnancy, i.e. positive urine pregnancy test

CONTACTS AND LOCATIONS:
Overall Officials: Antonios Likourezos, M.P.H., M.A., Study Director — Maimonides Medical Center
Locations (1):
- Genesis Fertility Center, Brooklyn, New York, United States